CLINICAL TRIAL: NCT02879565
Title: Families Expectations and Hope Raised by an Evaluation of Consciousness in Patients With an Unresponsive Wakefulness Syndrome
Brief Title: Families Expectations and Hope Raised by an Evaluation of Consciousness in Patients in a Vegetative State
Acronym: REVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Etablissement de rééducation fonctionnelle Les Salins de Bregille (Unknown); Etablissement de rééducation fonctionnelle, Bretégnier (Unknown); Hôpital Local de Bussang (Unknown); University of Franche-Comté (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: REVE
Record Dates: First submitted 2016-07-18; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Disorders of Consciousness; Qualitative Research; Ethics; Neuroimaging
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- qualitative and neuroimaging research (Other)
  Interventions: Other: Semi structured interviews + EEG exams

INTERVENTIONS:
Other: Semi structured interviews + EEG exams

SUMMARY:
Progress in resuscitation has increased the chances of survival after anoxic or traumatic brain injury. More and more patients with severe cerebral damages are resuscitated but upon awakening from coma, some patients remain in a state which cannot be qualified as conscious and is now known as an unresponsive wakefulness syndrome (UWS; formerly known as vegetative state). This condition can be transitory and evolve towards recovery, or remain chronic and lasting for years.

To improve the diagnosis of patients with disorders of consciousness, recent advances in brain imaging have led to the development of new methods of detecting awareness. In the absence of overt behavioral responses from these patients, imaging-based diagnostic methods have been first used to assess whether some cerebral areas were preserved in UWS patients and showed an activation of the primary sensory cortices in some UWS patients, whether it occurs at the auditory, visual or somatosensory level. Unavoidable technical and ethical issues are raised for clinicians before responding to such requests:

1. Is it technically possible to generalize neuroimaging protocols to all healthcare institutions?
2. Is it ethically acceptable to propose neuroimaging protocols without an accurate estimation of their psychological impact on families and caregivers?

The present study aims to understand and anticipate the technical and ethical issues related to an evaluation of consciousness with functional neuroimaging. How the evaluation of awareness in a patient affects the caregivers and family members will be investigated. By using qualitative research hopes and expectations will be clarified through the experiences of families, clinicians and nurses faced to this situation.

Will be included in this research professional caregivers and persons closely related to UWS patients:

* Family members or close circle visiting the patients on a regular basis
* Referring clinicians
* Nurses in charge of the patients' care

This prospective study uses qualitative, interview-based, research. Two key-moments are explored in succession to examine the impact of a neuroimaging evaluation of consciousness in institutionalized UWS patients:

* interviews of professional caregivers and families about their hopes concerning the evaluation of consciousness of UWS patients,
* interviews of professional caregivers and families about the impact of evaluating consciousness on their beliefs

ELIGIBILITY:
Inclusion Criteria:

* adult family members, clinicians, nurses (aged >18 years) closely related to UWS patients
* patients diagnosed as being in an UWS

Exclusion Criteria:

* patients in a minimally conscious state, in a locked-in-syndrome of akinetic mutism
* refusal of family members, clinicians or nurses to participate to the study
* family members considered by clinicians not to be capable of passing the interviews
* subjects aged < 18 years
* non french speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Perceptions of physicians and family members toward neuroimaging exams | day one
  semi-structured interviews before the neuroimaging exams

SECONDARY OUTCOMES:
Perceptions of physicians and family members of the neuroimaging exams results | day seven
  semi-structured interviews after the neuroimaging exams

CONTACTS AND LOCATIONS:
Overall Officials: Régis Aubry, Pr, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - Etablissement de rééducation fonctionnelle Les Salins de Bregille, Besançon
  - Etablissement de rééducation fonctionnelle Bretégnier, Héricourt